CLINICAL TRIAL: NCT01251640
Title: A Multi-center, Phase I/II Study of BAY86-9766 in Combination With Gemcitabine in Patients With Locally Advanced Inoperable or Metastatic Pancreatic Cancer
Brief Title: Combination With Gemcitabine in Advanced Pancreatic Cancer
Acronym: BAGPAC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14905; 2010-019588-12 (EudraCT Number)
Record Dates: First submitted 2010-11-08; First posted 2010-12-02 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreatic cancer,; MEK-inhibitor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-9766+Gemcitabine

INTERVENTIONS:
Drug: BAY86-9766+Gemcitabine — Phase I: 40 mg/day (20 mg twice daily), 60 mg/day (30 mg twice daily, 100 mg/day (50 mg bid) dependent on safety/tolerability Phase II: Recommended Phase II dose (RP2D) dependent on the results of the Phase I part of this study Route of administration: Oral, twice daily (bid) in combination with gemcitabine 1000 mg/m2 Intravenous infusion over 30 minutes weekly for seven out of eight weeks (Cycle 1); followed by 1000 mg/m2 Intravenous infusion over 30 minutes weekly for three out of four weeks (Cycle 2 and subsequent)

SUMMARY:
Open-label, uncontrolled, Phase I/II study to evaluate safety and efficacy of BAY86-9766 plus gemcitabine in locally advanced, unresectable or metastatic pancreatic cancer.

Phase I: Dose escalation study investigating 20, 30 and 50 mg BAY86-9766 plus gemcitabine (1000mg/m2); determination of maximum tolerated dose and recommended phase 2 dose.

Phase II: Determination of response (RECIST 1.1; primary endpoint). Secondary endpoints: response duration, disease control rate, time to progression, progression-free survival, overall survival, safety and tolerability.

Tumor assessments at Screening and than every 8 weeks.; Safety evaluations at Screening and weekly throughout the study; Safety follow-up visit 30 days after the last dose of study treatment; Survival follow up monthly for up to 8 month after LPFV.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years of age
* Histological or cytologically confirmed locally advanced, inoperable or metastatic pancreatic adenocarcinoma not amenable to curative radiotherapy or surgery
* Patients must have at least one uni-dimensional measurable lesion by CT or MRI according to RECIST, Version 1.1
* Resolution of all acute toxic effects of any prior local treatment to Common Terminology Criteria for Adverse Events (CTCAE) Grade </= 1
* Eastern Cooperative Oncology Group performance status (ECOG PS) </= 2
* Patient has cardiac function, within normal range, as measured by an echocardiogram

Exclusion Criteria:

* Known history of, or symptomatic metastatic brain or meningeal tumors
* History of cardiac disease
* Active clinically serious infections
* Clinically significant (ie. symptomatic) peripheral vascular disease
* Pregnant or lactating women; women of childbearing potential not employing adequate contraception
* Use of strong inhibitors or inducers of CYP3A4
* Prior systemic therapy for metastatic or locally advanced, unresectable pancreatic cancer, or other malignancy
* Previous gemcitabine or 5-fluorouracil (5-FU) given concurrently as radiosensitizers to radiation therapy in adjuvant intention if given within 6 months from start of study treatment
* Thrombotic or embolic events such within 6 months prior to start of study treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-02-11 (Actual); Study Completion 2013-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Dose Limiting Toxicities (DLT): Phase I | From randomization up to the first 8 weeks of therapy
Tumor Response (Adjudicated Blinded Read Assessment): Phase II | From start of treatment until 134 weeks assessed every 8 weeks

SECONDARY OUTCOMES:
Tumor Response: Investigator Assessment: Phase I | From start of treatment until 134 weeks assessed every 8 weeks
Disease Control (DC): Phase I | From start of treatment until 134 weeks assessed every 8 weeks
Disease Control (DC): Phase II | From start of treatment until 134 weeks assessed every 8 weeks
Duration of Response (DOR): Phase I | From start of treatment until 134 weeks assessed every 8 weeks
Duration of Response: Phase II | From start of treatment until 134 weeks assessed every 8 weeks
Time to Progression (TTP): Phase I | From start of treatment until 134 weeks assessed every 8 weeks
Time to Progression (TTP): Phase II | From start of treatment until 134 weeks assessed every 8 weeks
Progression-Free Survival (PFS): Phase I | From start of treatment until 134 weeks assessed every 8 weeks
Progression-Free Survival (PFS): Phase II | From start of treatment until 134 weeks assessed every 8 weeks
Overall Survival (OS): Phase I | From start of treatment until 134 weeks assessed every 8 weeks
Overall Survival (OS): Phase II | From start of treatment until 134 weeks assessed every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- United States (2):
  - Aurora, Colorado
  - Pittsfield, Massachusetts
- Belgium (2):
  - Bruxelles - Brussel
  - Edegem
- Czechia (2):
  - Brno
  - Olomouc
- Clermont-Ferrand, France
- Germany (5):
  - Heilbronn, Baden-Wurttemberg
  - München, Bavaria
  - Marburg, Hesse
  - Bochum, North Rhine-Westphalia
  - Berlin
- Italy (2):
  - Brescia, Lombardy
  - Ancona, The Marches
- Oslo, Norway
- Poland (3):
  - Bialystok
  - Gdansk
  - Warsaw
- London, United Kingdom

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/